CLINICAL TRIAL: NCT01882400
Title: Évaluation Multidimensionnelle de la réponse au Traitement de l'ostéoporose spontanée et Induite Par Les corticostéroïdes à l'Aide d'un Bisphosphonate à Administration Orale Chez Des Malades Porteurs d'Une Dystrophie Musculaire sévère.
Brief Title: Assessment of Response to Treatment of Osteoporosis With Oral Bisphosphonates in Patients With Muscular Dystrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilles Boire (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor-Investigator, Gilles Boire, Doctor Gilles Boire, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 01-12; Unrestricted grant (Other Grant/Funding Number: Procter&Gamble)
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Osteoporosis; Muscular Dystrophy; Cystic Fibrosis
Keywords: Osteoporosis; Severe muscular dystrophy; Cystic fibrosis
MeSH Terms: conditions — Osteoporosis; Muscular Dystrophies; Cystic Fibrosis | interventions — Risedronic Acid; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bisphosphonate treatment (Experimental): Add a weekly bisphosphonate to adequate doses of calcium and vitamin D supplements
  Interventions: Drug: Bisphosphonate treatment

INTERVENTIONS:
Drug: Bisphosphonate treatment — Treatment with Calcium, vitamin D and a weekly bisphosphonate. Comparison of bone mass, fracture rate, pain intensity and scoliosis progression before and after treatment
  Other Names: Risedronate; Alendronate

SUMMARY:
By supplying an adequate amount of calcium and vitamin D with the addition of weekly bisphosphonate, the investigators will be able to increase bone mass and decrease the incidence of fragility fractures in these children with muscular dystrophy.

The investigators think this treatment will also decrease the intensity of pain frequently present in these patients and slow the progression of scoliosis.

DETAILED DESCRIPTION:
Children with muscular dystrophy, as well as children with other chronic diseases (e.g. cystic fibrosis, chronic inflammatory arthritis) are at risk to develop fragility fractures both due to the disease itself and to drugs (mostly corticosteroids) used to treat the diseases.

In addition, children with muscular dystrophy frequently complain of diffuse pain making daily care more difficult and almost always develop structural scoliosis.

The objective of the present protocol is to offer these children a preventive treatment aimed at maintaining or increasing their bone mass. We also propose that maintaining bone mass will decrease fracture rates, as well as pain and the rate of progression of scoliosis.

Rigorous care to ensure adequate intake of calcium and vitamin D, as well as addition of a weekly bisphosphonate, are the central aspect of the project. In addition, we will monitor to avoid possible side-effects such as hypercalciuria and kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporosis or osteopenia
* Severe muscular dystrophy or cystic fibrosis
* May use corticosteroids

Exclusion Criteria:

* Inability to consent or to take drugs by mouth

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2001-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Increase in bone density according to osteodensitometry | Over 2 years of treatment
  comparing successive bone densitometry

SECONDARY OUTCOMES:
Decrease in bone pain | Over the first 2 years of treatment
  comparing reports of bone pain
Retardation of scoliosis development | Over the first 2 years of treatment
  computing how many patients had to have scoliosis surgery

OTHER OUTCOMES:
Side effects of treatment | Over 2 years
  Look for increases in kidney stones or hypercalciuria

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Boire, MD, MSc, Principal Investigator — CHUS and Université de Sherbrooke
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Jeffery TC, Chang AB, Conwell LS. Bisphosphonates for osteoporosis in people with cystic fibrosis. Cochrane Database Syst Rev. 2023 Jan 10;1(1):CD002010. doi: 10.1002/14651858.CD002010.pub5. PMID 36625789